CLINICAL TRIAL: NCT00311467
Title: Combined Treatment With Capecitabine and Immunotherapy Versus Immunotherapy Alone in Advanced Renal Cell Carcinoma: a Prospective, Randomized, Multi-center phaseIII-Trial
Brief Title: Combined Treatment With Capecitabine and Immunotherapy Versus Immunotherapy Alone in Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: no patient recruitment
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CECOG RCC 1.3.001
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Renal Cell Cancer
Keywords: renal cell cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Capecitabine; Interferons; Interleukins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capecitabine and Interferon (Active Comparator): Combined Chemo-Immunotherapy Chemotherapy: Mo-Fr Immunotherapy
  Interventions: Drug: Capecitabine, Interferon, Interleukin
- Interferon (Active Comparator): Patients randomized to group B will receive treatment according to the same treatment schedule and at the same dosages without capecitabine.
  Efficacy evaluations will be performed every 14 weeks of treatment in both groups
  Interventions: Drug: Capecitabine, Interferon, Interleukin

INTERVENTIONS:
Drug: Capecitabine, Interferon, Interleukin — Capecitabine orally from day 1 to 14 at a dose of 1000 mg/m2 twice daily every 21 days.
  Interferon-alpha subcutaneously on days 1 + 3 + 5 weeks 1 + 2 +6 + 7,11+12 at a dose of 6 MIU/d.
  Interleukin-2 subcutaneously on days 1 to 4 in weeks 3 + 4 +8 + 9,13+14 at a dose of 4.5 MIU/day.
  Group B
  Patients randomized to group B will receive treatment according to the same treatment schedule and at the same dosages without capecitabine.
  Efficacy evaluations will be performed every 14 weeks of treatment in both groups

SUMMARY:
Multi-center, prospective randomised phase III study evaluating capecitabine in combination with standard-immunotherapy versus standard-immunotherapy alone as first-line therapy in patients with metastatic renal cell carcinoma.

DETAILED DESCRIPTION:
Treatment plan Group A

Patients randomised to group A will receive treatment according to the following treatment schedule:

Group A: Combined Chemo-Immunotherapy Chemotherapy: Mo-Fr Immunotherapy

* Week 1:Capecitabine / Interferon;
* Week 2:Capecitabine / Interferon;
* Week 3:REST PERIOD / Interleukin;
* Week 4:Capecitabine / Interleukin;
* Week 5:Capecitabine / REST PERIOD;
* Week 6:REST PERIOD / Interferon;
* Week 7:Capecitabine / Interferon;
* Week 8:Capecitabine / Interleukin;
* Week 9:REST PERIOD / Interleukin;
* Week 10:Capecitabine / REST PERIOD;
* Week 11:Capecitabine / Interferon;
* Week 12:REST PERIOD / Interferon;
* Week 13:Capecitabine / Interleukin;
* Week 14:Capecitabine / Interleukin;

DOSAGES AND ROUTES OF ADMINISTRATION:

Capecitabine orally from day 1 to 14 at a dose of 1000 mg/m2 twice daily every 21 days.

Interferon-alpha subcutaneously on days 1 + 3 + 5 weeks 1 + 2 +6 + 7,11+12 at a dose of 6 MIU/d.

Interleukin-2 subcutaneously on days 1 to 4 in weeks 3 + 4 +8 + 9,13+14 at a dose of 4.5 MIU/day.

Group B

Patients randomized to group B will receive treatment according to the same treatment schedule and at the same dosages without capecitabine.

Efficacy evaluations will be performed every 14 weeks of treatment in both groups

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma (primary tumour or biopsy/surgery of metastases)
* Radiologically confirmed metastatic disease
* Surgically removed primary tumour so feasible (nephrectomy or nephron-sparing surgery as indicated)
* Karnofsky-Performance Status >70%
* Age 19-75 years
* Life expectancy of at least 3 months
* Adequate bone marrow function (i.e. white blood cell count above 3000/μL, platelet count above 75 000 /μL, hemoglobin above 9 mg/dl)
* Adequate organ function (i.e. serum creatinine, bilirubin and AST below 1.25 x the upper limit of the institutions' normal range)
* Negative pregnancy test for female patients
* Written informed consent

Exclusion Criteria:

* Age <19 or >75 years
* Karnofsky-Performance Status < 70%
* Untreated or uncontrolled brain metastases
* Second neoplasia
* Primary tumour surgically removable
* Solitary, surgically removable metastases
* Major concomitant diseases of the cardiovascular, respiratory or renal systems, as well as active systemic infections
* Severe renal disease or liver insufficiency or myeloid dysfunction (including patients with a history of a disease that is likely to interfere with the metabolism or excretion of the test medication)
* Other less common diseases as peptic ulcer disease, inflammatory bowel disease, autoimmune disease (severe known psoriasis, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis etc.)
* Drug addiction (including excessive alcohol consumption) within 1 year prior to study start.
* History of other conditions consistent with decompensated liver disease or other evidence of bleeding form esophageal varices.
* History of chronic hepatitis and immunsupressiva
* Known HIV Infection
* Evidence of allergy or hypersensitivity against recombinant Interferon alfa-2a or other components of preparation.
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease.
* Seizure disorders and /or compromised central nervous system function.
* History of evidence of severe retinopathy
* Patient unwilling or unable to give informed consent
* Pregnancy or breastfeeding

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2004-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary study objective is to investigate whether the addition of capecitabine to interferon-alpha-interleukin-2 based immunotherapy may improve progression free survival when compared to immunotherapy alone.

SECONDARY OUTCOMES:
The study's secondary objectives are to investigate differences in response rates, safety and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Schmidinger, Prof, Principal Investigator — Univ. Klinik f. Innere Med. I, Abt. Onkologie
Locations (1):
- Univ. Klinik f. Innere Medizin, Abt. Onkologie, Vienna, Austria

REFERENCES:
- See also: Related Info — http://www.cecog.org